CLINICAL TRIAL: NCT01477593
Title: Circumcision With a Novel Disposable Device in Chinese Children: a Hospital-based Randomized Controlled Trail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Feng Pan (Other)
Responsible Party: Sponsor-Investigator, Feng Pan, Clinical Attending Doctor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMU-124
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Circumcision
Keywords: circumcision, chinese children, pain
MeSH Terms: conditions — Pain | interventions — Circumcision, Male

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Experimental)
  Interventions: Procedure: circumcision with Shenghuan in Yan's method
- Group II (Active Comparator)
  Interventions: Procedure: circumcision with Shenghuan in Peng's method
- Group III (Active Comparator)
  Interventions: Procedure: conventional method with incision

INTERVENTIONS:
Procedure: circumcision with Shenghuan in Yan's method — The foreskin is first separated from the glans.Then the inner ring is placed between them and over the glans. After adjusting the position of inner ring to retain 0.5cm inner foreskin, the operator install the outer ring over the foreskin and combine them together. Removal of excess foreskin is then performed upon the device.
  Arms: Group I
Procedure: circumcision with Shenghuan in Peng's method — The foreskin is first separated from the glans. Then the inner ring is placed on the outer layer of foreskin. Next, the rim of the foreskin is clamped with blood vessel forceps at the 3, 6, 9 and 12 o'clock points. An urologist and an assistant each hold two clamps to widen the opening of the foreskin, and pull it over the inner ring. After the inner and outer layers of the foreskin and the frenulum are symmetrically positioned, the assistant install the outer ring over the foreskin and gently combine it together. Removal of excess foreskin is then performed below the device.
  Arms: Group II
Procedure: conventional method with incision — The procedure of conventional circumcision involve transection of the excess foreskin with reservation of 0.5cm inner foreskin, haemostasis by electrocautery and suture of skin edges with 4-0 absorption sutures.
  Arms: Group III

SUMMARY:
Circumcision, a removal of the foreskin, is performed commonly at any age in male worldwide. Globally over 25% of men are circumcised. In the Middle East, circumcision is even performed routinely in every male newborn. The benefits from it vastly outweigh the risks. Gradually, more and more Chinese male are willing to undergo it with themselves and their sons. But there are also some complications with circumcision, such as pain, edema, infection, and hemorrhage. Considering of that, physicians continually manage to improve their surgical methods and analgesic techniques.

In the study of Peng, a disposable minimally invasive circumcision anastomosis device named Shenghuan (China Wuhu Snnda Medical Treatment Application Technology Co. Ltd.) (ShD) was introduced to be applied in circumcision. And they concluded that method was quicker, safer and less pain than the conventional techniques of incision. In present study, we carry out a randomized controlled trail, using a different method as Peng introduced with this device in children's circumcision (Yan's), compared with the method as Peng used and the conventional technique in our hospital, and then observe the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children with phimosis or redundant prepuce

Exclusion Criteria:

* Children with genital tract infection or deformity,
* congenital diseases,
* hematological diseases,
* or other general diseases

Ages: 3 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
operation time | within operation

SECONDARY OUTCOMES:
pain score | within operation